CLINICAL TRIAL: NCT01745861
Title: Randomised Controlled Trial On The Effects Of Parenteral Fish Oil Emulsion In Patients With Severe Acute Pancreatitis
Brief Title: Effects Of Fish Oil Emulsion On Severe Acute Pancreatitis Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospitals, Leicester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SAP version 3 26-05-2011
Record Dates: First submitted 2012-11-13; First posted 2012-12-10 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2012-12

CONDITIONS: Assess Effect of Omega-3 Fish Oil in Patients With Severe Acute Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lipidem® (BBraun) (Active Comparator): Lipid emulsion containing medium chain triglycerides (MCT), long chain triglyceride (LCT) and Omega-3 fatty acid (fish oil)
  Interventions: Dietary Supplement: Lipidem (Omega-3 fish oil lipid emulsion)
- Lipofundin® MCT/LCT 20% (Placebo Comparator): Lipid emulsion containing medium and long chain triglycerides
  Interventions: Dietary Supplement: Lipofundin® MCT/LCT 20%

INTERVENTIONS:
Dietary Supplement: Lipidem (Omega-3 fish oil lipid emulsion) — Lipidem 200 mg/ml daily infusion for 7 days maximum
  Arms: Lipidem® (BBraun)
Dietary Supplement: Lipofundin® MCT/LCT 20% — Lipofundin® MCT/LCT 20% daily infusion for 7 days
  Arms: Lipofundin® MCT/LCT 20%

SUMMARY:
The incidence of acute pancreatitis in UK has risen sharply over the past 40 years. Recent reports suggest that 56.5 per 100 000 of the population will suffer from AP annually; this figure is more than double the highest previous estimated incidence. In the majority of patients the condition is mild, but about 25% of patients suffer a severe attack and between 30 and 50% of these patients dies. The usual cause of death is multiple organ failure secondary to systemic leukocyte activation (mainly neutrophils), accompanied by the systemic inflammatory response syndrome (SIRS).

Studies with omega-3 fish oil have shown to control inflammatory process and improve the outcome especially in hyperinflammatory conditions.

This research will look at the effects of supplementing omega-3 fish oil to patients with severe acute pancreatitis (severe inflammation of the pancreas).

Patients with severe acute pancreatitis will be prospectively and blindly randomised into either a study group who will receive (Lipidem, lipid emulsion contains essential fatty acids and omega-3 fish oil) or a control group that will receive (Lipofundin, lipid emulsion contains only essential fatty acids and no omega-3 fish oil). Normal and standard clinical care will be provided to all patients as per the national management guidelines. Each patient will receive either Lipidem or Lipofundin emulsions daily until they are deemed fit for discharge by their own medical team or for a maximum of SEVEN days.

The main aim of this study is to examine whether lipid emulsions enriched with omega-3 fish oil could improve the clinical outcome in patients with severe acute pancreatitis.

DETAILED DESCRIPTION:
This research project is designed to give lipid emulsion enriched with omega-3 fish oil to conscious adult patients with mental capacity to consent for themselves and with severe acute pancreatitis in Leicester General Hospital wards or units.

Potential participants with SAP will be identified by the patient's own team and referred to the researchers for consideration and eventual enrolling in the study. Unconscious patients or unable to consent for themselves will be EXCLUDED from the study.

Randomization:

Patients will be randomised to receive Lipidem 200 mg/ml OR Lipofundin MCT/LCT 20% lipid emulsion from random number tables. Randomization, blinding procedure (over labeling) will be conducted by an independent licensed pharmaceutical unit.

ELIGIBILITY:
Inclusion Criteria:

Conscious patients between age of 18-90 admitted to the Leicester General hospital with severe acute pancreatitis proven by:

1. compatible clinical features (abdominal pain with or without vomiting);
2. associated with elevated serum amylase levels (≥3 normal value) (≥300 iu/l);
3. one or more of the severity criteria as outlined in the Atlanta severity criteria or modified glasgow acute pancreatitis severity score ≥3

Exclusion Criteria:

* Patients unconscious or unable to consent.
* Patients under 18 years old or above 90 years old
* Hypersensitivity to fish, egg or soy protein or other active substances of the TPN.
* Uncontrolled hyperlipidaemia
* Severe primary blood coagulation disorder
* Acute pancreatitis accompanied with hyperlipidaemia
* Ketoacidosis
* Acute thromboembolic disease
* Severe liver failure
* Acute phase of myocardial infarction or stroke
* Pregnancy and lactation
* Severe renal failure without access to haemofiltration or dialysis

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Reduction of the CRP by 20% from the control group | Day 7 post infusion

SECONDARY OUTCOMES:
Progression in the Sequential Organ Failure Assessment (SOFA) Score | On days 1, 2, 3, 5 and 7 post infusion
Progression in the Multiple Organ Dysfunction Score (MODS) | On days 1, 2, 3, 5 and 7 post infusion
Progression in the Systemic Inflammatory Response Syndrome | On days 1, 2, 3, 5 and 7 post infusion
Progression in the inflammatory and anti-inflammatory mediators (IL-1RA, IL-10, IL-6, IL-18, TNF-a, ICAM-1, IL-10 etc...). | On days 1, 2, 3, 5 and 7 post infusion
Escalation of care to high dependency or intensive care unit and length of hospital stay | On days 1, 2, 3, 5 and 7 post infusion

CONTACTS AND LOCATIONS:
Overall Officials: Mr. Ashley Dennison, MD FRCS, Principal Investigator — Leicester General Hospital, University Hospitals of Leicester NHS Trust; Matthew Metcalfe, MD FRCS, Study Chair — Leicester General Hospital, University Hospitals of Leicester NHS Trust
Locations (1):
- Leicester General Hospital, University Hospitals of Leicester NHS Trust, Leicester, Leicestershire, United Kingdom

REFERENCES:
- [Background] Foitzik T, Eibl G, Schneider P, Wenger FA, Jacobi CA, Buhr HJ. Omega-3 fatty acid supplementation increases anti-inflammatory cytokines and attenuates systemic disease sequelae in experimental pancreatitis. JPEN J Parenter Enteral Nutr. 2002 Nov-Dec;26(6):351-6. doi: 10.1177/0148607102026006351. PMID 12405646
- [Background] Morlion BJ, Torwesten E, Lessire H, Sturm G, Peskar BM, Furst P, Puchstein C. The effect of parenteral fish oil on leukocyte membrane fatty acid composition and leukotriene-synthesizing capacity in patients with postoperative trauma. Metabolism. 1996 Oct;45(10):1208-13. doi: 10.1016/s0026-0495(96)90237-1. PMID 8843174
- [Background] Hardman WE. (n-3) fatty acids and cancer therapy. J Nutr. 2004 Dec;134(12 Suppl):3427S-3430S. doi: 10.1093/jn/134.12.3427S. PMID 15570049
- [Background] Roulet M, Frascarolo P, Pilet M, Chapuis G. Effects of intravenously infused fish oil on platelet fatty acid phospholipid composition and on platelet function in postoperative trauma. JPEN J Parenter Enteral Nutr. 1997 Sep-Oct;21(5):296-301. doi: 10.1177/0148607197021005296. PMID 9323693
- [Background] Serhan CN, Clish CB, Brannon J, Colgan SP, Chiang N, Gronert K. Novel functional sets of lipid-derived mediators with antiinflammatory actions generated from omega-3 fatty acids via cyclooxygenase 2-nonsteroidal antiinflammatory drugs and transcellular processing. J Exp Med. 2000 Oct 16;192(8):1197-204. doi: 10.1084/jem.192.8.1197. PMID 11034610
- [Background] Lee TH, Hoover RL, Williams JD, Sperling RI, Ravalese J 3rd, Spur BW, Robinson DR, Corey EJ, Lewis RA, Austen KF. Effect of dietary enrichment with eicosapentaenoic and docosahexaenoic acids on in vitro neutrophil and monocyte leukotriene generation and neutrophil function. N Engl J Med. 1985 May 9;312(19):1217-24. doi: 10.1056/NEJM198505093121903. PMID 2985986
- [Derived] Al-Leswas D, Eltweri AM, Chung WY, Arshad A, Stephenson JA, Al-Taan O, Pollard C, Fisk HL, Calder PC, Garcea G, Metcalfe MS, Dennison AR. Intravenous omega-3 fatty acids are associated with better clinical outcome and less inflammation in patients with predicted severe acute pancreatitis: A randomised double blind controlled trial. Clin Nutr. 2020 Sep;39(9):2711-2719. doi: 10.1016/j.clnu.2018.04.003. Epub 2018 Apr 27. PMID 32921364